CLINICAL TRIAL: NCT00526773
Title: Enhancing Heart Failure Self-Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Angela DiSabatino, RN, MS, Manager, Cardiovascular Clinical Trials Program, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCC27020
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Heart Failure
Keywords: motivational therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Telephone management plus a motivational intervention
  Interventions: Other: telephone management plus a motivational intervention
- 2 (Other): Telephone management with standard patient education
  Interventions: Other: telephone management with standard patient education

INTERVENTIONS:
Other: telephone management plus a motivational intervention — heart failure intervention
  Arms: 1
Other: telephone management with standard patient education — heart failure intervention
  Arms: 2

SUMMARY:
To test the effectiveness of a motivational intervention compared with standard patient education in improving economic and clinical outcomes in patients enrolled in an existing heart failure (HF) disease management program.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure, hospitalized for heart failure or hospitalized for heart failure within the past 30 days, speak and read English

Exclusion Criteria:

* Severe renal failure requiring dialysis, HIV-AIDS, psychosis, uncorrected hearing loss

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To test the effectiveness of a motivational intervention compared with standard patient education in improving economic and clinical outcomes in patients enrolled in HF disease management. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Reigel, DNSc, RN, CS, FAAN, Principal Investigator — University of Pennsylvania
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States